CLINICAL TRIAL: NCT01548040
Title: A Randomised Controlled Study To Compare the Effects of a Standard Therapy Protocol With a 12-week Peri-Operative Program of Kneehab XP Compared to a Control Treatment in Patients Undergoing Total Knee Replacement
Brief Title: Controlled Study of Kneehab XP for Patients Undergoing Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theragen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00012744
Record Dates: First submitted 2012-02-16; First posted 2012-03-08 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: Total Knee Replacement
Keywords: NMES; Muscle; strength; TKA; Focus to show shorter muscle recovery after Knee operation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- quadriceps NMES using Kneehab XP (Experimental): All subjects in the treatment group will receive quadriceps Neuro Muscular Electrical Stimulation (NMES) using Kneehab XP on the affected leg, 20 minutes, twice per day, 5 days a week. Subjects will begin use of the device at 6 weeks pre-operatively and continue through 6 weeks post-operatively.group will also complete the standard TKA post-surgery rehabilitation program used at the Hawkins Foundation
  Interventions: Device: Kneehab XP
- quadriceps TENS (Sham Comparator): The sham device will look identical to the Kneehab XP device. All subjects in the control group will receive quadriceps Transcutaneous Electrical Nerve Stimulation (TENS) at a minimal sensory input using Kneehab XP on the affected leg, 20 minutes, twice per days, 5 days a week. Subjects will begin use of the device at 6 weeks pre-operatively and continue through 6 weeks post-operatively.group will also complete the standard TKA post-surgery rehabilitation program used at the Hawkins Foundation
  Interventions: Device: Quadriceps TENS

INTERVENTIONS:
Device: Kneehab XP — NMES using Kneehab XP on the affected leg,20 minutes, twice per day, 5 days a week. Subjects will begin use of the device at 6 weeks pre-operatively and continue through 6 weeks post-operatively
  Arms: quadriceps NMES using Kneehab XP
Device: Quadriceps TENS — on the affected leg, 20 minutes, twice per days, 5 days a week. Subjects will begin use of the device at 6 weeks pre-operatively and continue through 6 weeks post-operatively.
  Arms: quadriceps TENS

SUMMARY:
The study is a prospective, randomized, double-blind sham study of TKA patients who receive a standard peri-operative treatment program plus Kneehab XP versus a standard peri-operative treatment program plus a sham device.

DETAILED DESCRIPTION:
The study is a double-blind randomized controlled clinical trial of approximately 118 patients (males and females) who are at least 40 years of age, who are scheduled for Total Knee Arthroplasty (TKA) surgery will be randomized into 1) a treatment group who receive Kneehab XP and a standard rehabilitation program and 2) a control group who receive only a sham device and a standard rehabilitation program. Patients are tracked for measures of function, pain, quality of life, physical performance and acceptable states status at 6 weeks and 1 week before surgery and 3, 6, 12, and 52 weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are scheduled for Total Knee Replacement surgery with the Smith and Nephew Visionaire prosthesis and the anterior surgical approach.
* Individuals who are at least 40 years of age.
* Individuals with a body mass index (BMI) <40 kg/ m2
* Individuals who are walking independently with or without assistive devices.
* Individuals with a Short Performance Battery Score greater than 7.
* Must be able and willing to complete all study assessments and to be followed for the full course of the study.
* Must be able to read, write and follow instructions in English.
* Must be able and willing to provide informed consent.
* Must be willing and able to attend the additional pre-operative assessment.

Exclusion Criteria:

* Individuals with a history of foot and/or ankle pathology.
* Individuals with a history of tibial or femoral fractures.
* Individuals with a history of any underlying neurological conditions.
* Individuals with physical conditions which would make them unable to perform study procedures.
* Individuals with a total hip replacement.
* Individuals undergoing revision TKA of the same operated leg.
* Individuals who are pregnant.
* Individuals diagnosed with a medical condition that would contraindicate treatment with the product, e.g. skin lesions at electrode site.
* Individuals with an active implanted medical device (i.e. pacemaker, pump)
* Individuals with a history of stroke
* Individuals with a history of neurological disorder that affects lower extremity function (stroke, peripheral neuropathy, Parkinson's disease, multiple sclerosis, etc.)
* Individuals with a diagnosis of inflammatory arthritis (Rheumatoid arthritis, gout or psoriatic arthritis).
* Individuals with muscle diseases (i.e. muscular dystrophy)
* Individuals with visible skin injury or disease on their legs.
* Individuals who have been committed to an institution by virtue of an order issued either by the courts or by an authority.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Burnikel, Principal Investigator — Hawkins Foundation
Locations (1):
- Hawkins Foundation, Greenville, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Quadriceps NMES Using Kneehab XP: All subjects in the treatment group will receive quadriceps NMES using Kneehab XP on the affected leg, 20 minutes, twice per day, 5 days a week. Subjects will begin use of the device at 6 weeks pre-operatively and continue through 6 weeks post-operatively.group will also complete the standard TKA post-surgery rehabilitation program used at the Hawkins Foundation
  Kneehab XP: NMES using Kneehab XP on the affected leg,20 minutes, twice per day, 5 days a week. Subjects will begin use of the device at 6 weeks pre-operatively and continue through 6 weeks post-operatively
- Quadriceps TENS: The sham device will look identical to the Kneehab XP device. All subjects in the control group will receive quadriceps TENS (at a minimal sensory input) using Kneehab XP on the affected leg, 20 minutes, twice per days, 5 days a week. Subjects will begin use of the device at 6 weeks pre-operatively and continue through 6 weeks post-operatively.group will also complete the standard TKA post-surgery rehabilitation program used at the Hawkins Foundation
  quadriceps TENS (at a minimal sensory input) using Kneehab XP: on the affected leg, 20 minutes, twice per days, 5 days a week. Subjects will begin use of the device at 6 weeks pre-operatively and continue through 6 weeks post-operatively.
Period: Overall Study
Arm/Group | Quadriceps NMES Using Kneehab XP | Quadriceps TENS
Started | 56 | 55
Completed | 43 | 45
Not Completed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadriceps NMES Using Kneehab XP | Quadriceps TENS | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.23) | 64.5 (10.23) | 64.8 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 24 | 23 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 56 | 55 | 111
Smoking Status [Count of Participants; unit: Participants]
  Current | 3 | 1 | 4
  Non | 36 | 34 | 70
  Ex | 17 | 20 | 37
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 30.0 (5.03) | 29.4 (5.23) | 29.7 (5.11)

OUTCOME MEASURES:

1. Primary Outcome: Isometric Strength Test
Description: To determine the efficacy of Kneehab XP in promoting early quadriceps strength improvement (measured as the difference between the baseline time point and the 6 week post-operative time point) when compared to a control group in patients undergoing total knee arthroplasty. Isometric strength was measured using a Biodex Isokinetic Dynamometer machine on patients seated and secured to a chair and who performed 3 maximal voluntary contractions (MVC) for which the maximal torque is measured and a mean taken of 3 consecutive MVC's.
Time Frame: measured at the 6 week post-operative time point
Measure: Mean (Standard Deviation); unit: Newton-metres
Arm/Group | Quadriceps NMES Using Kneehab XP | Quadriceps TENS
Number analyzed (Participants) | 56 | 55
Newton-metres | -21.9 (21.74) | -31.9 (28.43)

2. Secondary Outcome: Percentage of Patients With Positive PASS
Description: To determine whether Kneehab XP leads to earlier recovery (measured at the 6 week post-operative time point) when compared to a control group in patients undergoing total knee arthroplasty. Patient Acceptable Symptom State (PASS) is a yes/no answer to a specifically stated question about the patients satisfaction with their state. For clarity, Positive PASS implies that the answer that is given is Positive i.e. Yes
Time Frame: measured at the 6 week post-operative time point
Measure: Number; unit: % of participants
Arm/Group | Quadriceps NMES Using Kneehab XP | Quadriceps TENS
Number analyzed (Participants) | 56 | 55
% of participants
  Baseline | 25.0 | 16.4
  6 week post-surgery | 73.5 | 61.2

3. Other Pre Specified Outcome: Physical Therapy Sessions
Description: Change in patient functional measures and number of therapy sessions required.
Time Frame: 1 wk pre-operatively, 3,6,12,52 week post operatively
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Questionnaires
Description: Change in scores in patient outcome measures, functional measures and physical performance measures
Time Frame: 1 wk pre-operatively, 3,6,12,52 week post operatively
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Range of Motion
Description: Change in scores of functional and physical performance scores
Time Frame: 1 wk pre-operatively, 3,6,12,52 week post operatively
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Timed to Get up and go
Description: Change in scores of physical performance measures
Time Frame: 1 wk pre-operatively, 3,6,12,52 week post operatively
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Stair Climb Test
Description: Change in scores of physical performance measures
Time Frame: 1 wk pre-operatively, 3,6,12,52 week post operatively
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Visual Analogue Scales (VAS)
Description: Pain change score in VAS from baseline to week 6 post-surgery
Time Frame: 1 wk pre-operatively,3,6,12 and 52 post operatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Quadriceps NMES Using Kneehab XP | Quadriceps TENS
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55
Other Adverse Events (participants affected / at risk) | 7/56 | 0/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadriceps NMES Using Kneehab XP (N=56) | Quadriceps TENS (N=55)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pain (General disorders) | 4 (4) | 0 (0) — Mild pain associated with device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No